CLINICAL TRIAL: NCT03516552
Title: Comparison and Analysis of Blood Loss Formulas
Status: Completed | Type: Observational
Sponsor: Hospital Clinic of Barcelona (Other)
Responsible Party: Principal Investigator, Sebastian Jaramillo, MD, Hospital Clinic of Barcelona
Other Study IDs: 2016/0906
Record Dates: First submitted 2018-04-15; First posted 2018-05-04 (Actual); Last update posted 2019-08-07 (Actual); Status verified 2019-08

CONDITIONS: Blood Loss
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Hemoglobin content on blood loss: Hemoglobin content on blood loss, to assess ratio hemoglobin/volume.

SUMMARY:
Although it has been pointed that estimates are significantly inexact and different from each other, the actual accuracy of them has not been properly investigated and compared.

ELIGIBILITY:
Inclusion Criteria:

- Adults 18 - 90 yrs.

Exclusion Criteria:

* Suspected or confirmed coagulopathy (including current treatment with anticoagulants or antiplatelet agents).
* Surgical blood loss volume < 200 ml.
* Requirement for surgical gauzes during surgery, including conversion to open surgical techniques.
* Transfusion of red blood cells (RBCs) during the perioperative period.
* Significant postoperative bleeding (> 50 ml in surgical drains) or any other type of significant blood loss.
* Fluid infusions or vasoactive drugs after the first 24 postoperative hours.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients electively scheduled for laparoscopic surgery.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-08-10 (Actual)

PRIMARY OUTCOMES:
Differences on blood loss estimation. | 72 hours.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clinic de Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No